CLINICAL TRIAL: NCT05167253
Title: A Phase I, Open-label Study to Evaluate the Ability of UB-612 Vaccine to Boost Immunity of Heterologous COVID-19 Vaccines
Brief Title: A Study to Evaluate the Ability of UB-612 COVID-19 Vaccine to Boost Immunity of Heterologous COVID-19 Vaccines.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Regulatory issues raised by the regulatory authority in Taiwan.
Sponsor: United Biomedical Inc., Asia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V-125
Record Dates: First submitted 2021-12-16; First posted 2021-12-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — UB-612 COVID-19 vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UB-612 100 μg, 0.5 mL (Experimental): All subjects will be enrolled to receive one dose of 100 μg UB-612 vaccine
  Interventions: Biological: UB-612

INTERVENTIONS:
Biological: UB-612 — UB-612 includes a designer S1-RBD-sFc fusion protein formulated with designer Th and CTL epitope peptides selected from immunodominant M, S2 and N regions known to bind to human MHC I and II.

SUMMARY:
This is a study to evaluate the ability of UB-612 vaccine to boost immunity of subjects who previously received two doses of AstraZeneca COVID-19 vaccine (ChAdOx1-S) with an 8-16 week interval between first and second doses.

DETAILED DESCRIPTION:
This is a phase I, open-label clinical study to evaluate the ability of UB-612 vaccine to boost immunity of subjects who previously received two doses of AstraZeneca COVID-19 vaccine (ChAdOx1-S) with an 8-16 week interval between first and second doses.

This study will enroll approximately 30 subjects aged 20 to 55 years. The previous COVID-19 vaccine series will have been completed at least six months before study enrollment. Both sexes should be evenly distributed in subjects.

Subjects will be enrolled to receive one dose of 100 μg UB-612 vaccine at Day 1. The subjects will come to the clinics at Visit 1 (screening, Day -28 to -1), Visit 2 (Day 1, vaccination), Visit 3 (Day 15, 14 days after vaccination), Visit 4 (Day 29, 28 days after vaccination), Visit 5 (Day 169, 6 months after vaccination) and will receive phone calls at 7 days after vaccination for safety check.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female between the age of 20 and 55 years at time of enrolment.
* Fully vaccinated with two injections of AstraZeneca COVID-19 vaccine (ChAdOx1-S) with an 8-16 week interval between first and second doses. The second dose of AstraZeneca COVID-19 vaccine (ChAdOx1-S) must have been administered more than six (6) months from study Day 1. The CDC COVID-19 Vaccination Record Card or appropriate documentation (e.g., medical records) will be required for documentation.
* Women of childbearing potential and men must agree to practice medically effective contraception from vaccination until 30 days after the vaccination.
* Participant or the participant's legal representative must understand the procedures of the study and is willing to sign the Informed Consent Form (ICF).
* Able to understand and agrees to comply with all study procedures and be available for all study visits.
* Must be able to read, understand, and complete the protocol-required questionnaires and/or diary.
* Negative serological test for Hepatitis B surface antigen (HBsAg), HCV RNA and HIV antibody
* Negative results of SARS-CoV-2 N protein IgG ELISA
* Negative result of RT-PCR screening of nasopharyngeal or throat swabs for SARS-CoV-2.
* Ear temperature ≤ 38.0°C.
* Indexes of hematology, biochemistry and immunology laboratory tests are within the normal ranges, or not clinically significant as judged by investigators

Exclusion Criteria:

* History of anaphylaxis, urticarial, or other significant adverse reaction requiring medical intervention after receipt of a vaccine.
* Female who is pregnant or positive in pregnancy test at screening or just prior to vaccination administration or plans to become pregnant from the time of study vaccination through 30 days after the administration of the study vaccine.
* Female who is breast-feeding or plans to breastfeed from the time of the study vaccination through 30 days after the administration of the study vaccine.
* Investigational non-coronavirus vaccines: previous receipt of an investigational vaccine (non-coronavirus) within 1 year before the planned administration of study vaccine.
* Prior administration of attenuated, nucleic acid (mRNA or DNA) or vectored vaccines in last 1 month before the study vaccine or expectation of such vaccines in the month after the study vaccine.
* Prior administration of subunit vaccine or inactivated vaccine in last 14 days before the study vaccine or expectation of receipt of such vaccines in the 14 days after the study vaccine.
* Judged by the investigator on the basis of evidence or medical history, immunosuppressive or immunodeficient state, autoimmune diseases, chronic kidney disease (with dialysis), asplenia, or recurrent severe infections.
* Prior chronic administration of immunosuppressant or corticosteroids, cytotoxic treatment in last 6 months before the study vaccination.
* Receipt of short-term systemic corticosteroids. Study intervention administration should be delayed until systemic corticosteroid use has been discontinued for at least 28 days. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Has received systemic immunoglobulins or blood products within 4 months prior to enrollment.
* Loss or donation of blood over 500 mL within 3 months prior to screening visit or intention to donate blood or blood products for transfusion during the study.
* Participants who received specific anti-SARS-CoV-2 monoclonal antibody products at any time.
* Subjects who take part in another clinical study and are currently receiving or received any investigational intervention within 12 weeks prior to the day of informed consent.
* Platelet disorder or other bleeding disorder may cause injection contraindication.
* Any acute illness, as determined by the study investigator 3 days before vaccination.
* Judged by the investigator on the basis of evidence or medical history, participants with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies) will be excluded.
* History of malignancy within 5 years prior to screening visit, except basal cell carcinoma of the skin and cervical carcinoma in situ.
* Known history of SARS, MERS or SARS-CoV-2 infection.
* Alcoholism or substance abuser.
* Behavioral, cognitive, or psychiatric disease that, in the opinion of investigators, affects the participant's ability to understand and cooperate with all study protocol requirements.
* Employees at the investigator's site, of the Sponsor or the contract research organization (CRO) directly involved in the conduct of the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | within 7 days after vaccination
  * Local solicited adverse events
  * Systemic solicited adverse events
  * Skin allergic reactions
Safety and tolerability | 28 days after vaccination
  • Unsolicited adverse events
Immunogenicity | 14 days after vaccination
  • Geometric mean titers (GMT) of neutralizing antibody against SARS-CoV-2 wild type
Immunogenicity | 14 days after vaccination
  • Seroconversion rate (SCR) of neutralizing antibody against SARS-CoV-2 wild type
Immunogenicity | 14 days after vaccination
  • Geometric mean fold increase (GMFI) of neutralizing antibody against SARS-CoV-2 wild type

SECONDARY OUTCOMES:
Safety | Day 1
  * Adverse events)
  * AE of special interest
  * Vaccine-associated enhanced disease
  * Serious adverse events
  * Medically attended adverse events
Safety | 14 days after vaccination
  * Adverse events)
  * AE of special interest
  * Vaccine-associated enhanced disease
  * Serious adverse events
  * Medically attended adverse events
Safety | 28 days after vaccination
  * Adverse events)
  * AE of special interest
  * Vaccine-associated enhanced disease
  * Serious adverse events
  * Medically attended adverse events
Safety | 6 months after vaccination
  * Adverse events)
  * AE of special interest
  * Vaccine-associated enhanced disease
  * Serious adverse events
  * Medically attended adverse events
Evaluation of safety of hematology and biochemistry | Pre-vaccination
  Change of safety laboratory measurement from pre-vaccination
Immunogenicity | 14 days after vaccination
  • GMT of neutralizing antibody against SARS-CoV-2 wild type, antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 14 days after vaccination
  • SCR of neutralizing antibody against SARS-CoV-2 wild type, , antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 14 days after vaccination
  • GMFI of neutralizing antibody against SARS-CoV-2 wild type, , antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 28 days after vaccination
  • GMT of neutralizing antibody against SARS-CoV-2 wild type, antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 28 days after vaccination
  • SCR of neutralizing antibody against SARS-CoV-2 wild type, antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 28 days after vaccination
  • GMFI of neutralizing antibody against SARS-CoV-2 wild type, , antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 6 months after vaccination
  • GMT of neutralizing antibody against SARS-CoV-2 wild type, , antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 6 months after vaccination
  • SCR of neutralizing antibody against SARS-CoV-2 wild type, , antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 6 months after vaccination
  • GMFI of neutralizing antibody against SARS-CoV-2 wild type, , antigen-specific antibody titers (anti-S1-RBD), S1-RBD:ACE2 binding inhibition antibody
Immunogenicity | 14 days after vaccination
  • GMT of neutralizing antibody titers against SARS-CoV-2 variant
Immunogenicity | 14 days after vaccination
  • SCR of neutralizing antibody titers against SARS-CoV-2 variant
Immunogenicity | 14 days after vaccination
  • GMFI of neutralizing antibody titers against SARS-CoV-2 variant
Immunogenicity | 14 days after vaccination
  • Reduction fold of GMT compared with neutralizing antibody titers against SARS-CoV-2 wild type
Immunogenicity | 28 days after vaccination
  • GMT of neutralizing antibody titers against SARS-CoV-2 variant
Immunogenicity | 28 days after vaccination
  • SCR of neutralizing antibody titers against SARS-CoV-2 variant
Immunogenicity | 28 days after vaccination
  • GMFI of neutralizing antibody titers against SARS-CoV-2 variant
Immunogenicity | 28 days after vaccination
  • Reduction fold of GMT compared with neutralizing antibody titers against SARS-CoV-2 wild type
Immunogenicity | Day 1
  • T cell responses
Immunogenicity | 14 days after vaccination
  • T cell responses

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Yi Wang, Ph.D., Study Chair — United Biomedical Inc., Asia